CLINICAL TRIAL: NCT06492993
Title: Community Health Navigator Program to Promote Cancer Screenings Among Deaf, Deafblind, and Hard of Hearing Adults Who Use American Sign Language
Brief Title: Community Health Navigator Program to Promote Cancer Screenings Among DDBHH People
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gallaudet University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: CDHE
Record Dates: First submitted 2024-06-27; First posted 2024-07-09 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Deafness
MeSH Terms: conditions — Neoplasms; Deafness | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): CHN provides educational sessions with patients at time points.
  Interventions: Other: Education
- Standard of Care (No Intervention): Standard of care to inform participant about the screening recommendations and check ins.

INTERVENTIONS:
Other: Education — The CHN meets with DDBHH participant over sessions to provide navigation support through the cancer screening process.
  Arms: Intervention

SUMMARY:
Intervention to promote cancer screenings among deaf, deafblind, and hard of hearing participants who have not received screening within the recommended guideline.

DETAILED DESCRIPTION:
Study hypothesizes that the intervention that involves utilization of a DDBHH CHN will result in (i) DDBHH patients demonstrating greater adherence to screening compared to DDBHH patients who were assigned to the standard of care group , and (ii) higher patient-physician communication rating by DDBHH patients compared to DDBHH patients who were assigned to the standard of care group. Bilingual ASL-English measures (e.g., sociodemographics, cancer knowledge, patient-physician communication) will be administered to the participant at baseline data collection and again after the final data collection or by 11 months for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form

Stated willingness to comply with all study procedures and lifestyle considerations (see Section 5.3, Lifestyle Considerations) and availability for the duration of the study

Male or female at birth age 45-80yo or female at birth age 45-80yo; age-eligible according to screening criteria

Self-reported diagnosis of bilateral hearing loss at birth or prior to 13 years old (defined as "early deafness") and use ASL

Willingness to adhere to the CHN clinical trial regimen

Willingness to provide cancer screening verification documentation; this will be reviewed during the informed consent procedure

Access to necessary resources to support video-based communication

Non-adherent to one or more cancer screening guidelines for breast, lung, prostate, colon, cervical cancers will be those who reported not having had the appropriate recommended screenings within the past year to cancer screening questions in the HINTS-ASL survey

Exclusion Criteria:

* Presence of full ability to hear in one or both ears beyond 13 years of age

Younger or older than the age cutoff for the recommended cancer screening

Not capable of independently conducting the activities of daily living

In compliance with age- or risk-specific screening at the time of evaluation for study eligibility

Are currently undergoing cancer treatment or being evaluated for the presence of cancer at the time of evaluation for study eligibility

Will be engaged in more than 21 consecutive days of travel during the eleven-month study window

Knows other participants at baseline

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are adherent to cancer screening | 9 months
  Completion of at least one recommended cancer screening as measured by documentation of the actual screening

SECONDARY OUTCOMES:
Percent of participants who demonstrate high cancer knowledge and high perceived patient centered care | 9 months
  Positive change in patient-physician communication and cancer knowledge from baseline to closeout as defined by the participating patient.

CONTACTS AND LOCATIONS:
Overall Officials: Poorna Kushalnagar, Principal Investigator — Gallaudet University
Locations (1):
- Gallaudet University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kushalnagar P, Rao SR, Bergeron E, Valdez R, Wang R, Kushalnagar RS, Sadler GR. Using American Sign Language-Fluent Community Health Navigators to Advance Cancer Screening Adherence through Videoconferencing With Deaf, Deafblind, and Hard of Hearing Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 9;14:e65078. doi: 10.2196/65078. PMID 40925603